CLINICAL TRIAL: NCT01769612
Title: Evaluation of a Diagnostic Device, CL Detect Rapid Test, for the Diagnosis of Cutaneous Leishmaniasis in Tunisia
Brief Title: Evaluation of a Rapid Diagnostic Device, CL Detect, for the Diagnosis of Cutaneous Leishmaniasis in Tunisia
Acronym: CL Detect™
Status: Completed | Type: Observational
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: InBios International, Inc. (Industry); Institut Pasteur of Tunis, Tunisia (Unknown)
Responsible Party: Sponsor
Other Study IDs: S-12-14; A-15174.2b (Other: HRPO); K141341 (Other: Other)
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-04

CONDITIONS: Skin Diseases, Parasitic
Keywords: Leishmaniasis, Leishmania
MeSH Terms: conditions — Skin Diseases, Parasitic; Leishmaniasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- CL Detect Rapid Test and Microsopy Samples: Samples taken to be evaluated in the CL Detect and Microscopy assays
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
The purpose of the study is to evaluate the sensitivity and specificity of CL Detect, in subjects with suspected CL in Tunisia.

DETAILED DESCRIPTION:
Subjects were selected based on clinical appearance of the skin lesion characteristics of cutaneous leishmaniasis (CL). Study compared the CL Detect Rapid Test vs microscopic identification of Leishmania amastigotes in a stained lesion sample. Two diagnostic samples were collected from the subjects lesion in the following order: 1) obtained with a dental broach for use with the CL Detect Rapid Test and 2) a second sample was obtained by scraping for use in the microscopic identification of amastigotes. Samples were analyzed by microscopy and CL Detect Repaid Test by different operators who evaluated each sample independently blinded to the other assay result.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and generally healthy
* Subject able to give written informed consent
* Subject has a lesion suspicious for leishmaniasis that satisfies the following criteria for an index lesion:

  * less than 4 months in age
  * primarily ulcerative, ie not purely verrucous or nodular, and does not have clear clinical evidence of cellulitis
  * in a location suitable for collecting samples by dental broach, scraping, and aspiration
* In the opinion of the investigator, the subject is capable of understanding and complying with the protocol

Exclusion Criteria:

• Received treatment for leishmaniasis within the last 2 months prior to signing consent, with the exception of mercurochrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afif Ben Salah, MD PhD, Principal Investigator — Institut Pasteur de Tunis
Locations (2):
- Tunisia (2):
  - Primary Health Clinic, Gafsa, Gafsa Governorate
  - Primary Health Clinics, Sidi Bouzid, Sidi Bouzid Governorate

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 168 subjects were enrolled in the regions of Sidi Bouzid and Gafsa, Tunisia
Groups:
- CL Detect Rapid Test and Microsopy Samples: Samples taken to be evaluated in the CL Detect and Microscopy assays
  No Intervention
Period: Overall Study
Arm/Group | CL Detect Rapid Test and Microsopy Samples
Started | 168
Completed | 168
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CL Detect Rapid Test and Microsopy Samples
Number analyzed (Participants) | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  North African | 168
Region of Enrollment [Number; unit: participants]
  Tunisia | 168
Lesion Age [Mean (Standard Deviation); unit: days] | 36.2 (22.6)
Lesion Characteristics [Count of Participants; unit: Participants]
  Ulcerated | 168
  Nobular | 0
  Secondary bacterial infection | 74
Lesion Location [Count of Participants; unit: Participants]
  Abdomen | 0
  Arm | 55
  Back of head | 1
  Face | 4
  Foot | 35
  Hand | 14
  Leg | 59

OUTCOME MEASURES:

1. Primary Outcome: Positive Result Comparison: CL Detect Rapid Test With Microscopy and Culture Results
Description: Comparison of CL Detect Rapid Test positive results with Microscopy and Culture results.
  Note: only data where results for all three methods were available were included in the analysis.
Time Frame: within 1 hour after taking samples
Measure: Count of Participants; unit: Participants
Groups:
- CL Detect Rapid Test: Data for CL Detect Rapid Test
- Microscopy: Data for Micrscopy
- Culture: Data for Culture results
Arm/Group | CL Detect Rapid Test | Microscopy | Culture
Number analyzed (Participants) | 147 | 147 | 147
Participants | 147 | 144 | 96

ADVERSE EVENTS:
Time Frame: 48 hours after taking of samples
Arm/Group | CL Detect Rapid Test and Microsopy Samples
All-Cause Mortality (participants affected / at risk) | 0/168
Serious Adverse Events (participants affected / at risk) | 0/168
Other Adverse Events (participants affected / at risk) | 0/168

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No